CLINICAL TRIAL: NCT04452773
Title: Double-blind, Randomized, Placebo-Controlled Clinical Trial to Evaluate the Efficacy of the Manremyc® Food Supplement to Prevent SARS-CoV-2 Infection
Brief Title: Clinical Trial to Evaluate the Efficacy of Food Supplement Manremyc® Against SARS- COV-2 Infection (COVID-19) in Healthcare Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Reig Jofre Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MANRECOVID19
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manremyc (Experimental): Participants will receive daily oral administration of a capsule of Manremyc for 14 days in the morning with breakfast
  Interventions: Dietary Supplement: Manremyc
- Placebo (Placebo Comparator): Participants will receive daily oral administration of a capsule of Placebo for 14 days in the morning with breakfast
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Manremyc — Manremyc is composed by 10E5 heat-inactivated Mycobacterium s. manresensis bacilli
  Arms: Manremyc
Dietary Supplement: Placebo — Same excipients than active arm without bacilli.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of Manremyc® food supplement for reduce the incidence of SARS-CoV-2 infection in a high risk population, as healthcare workers.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the Informed Consent before initiating the selection procedures.
2. Health system workers working in contact with subjects potentially infected with SARS-CoV-2.
3. People ≥ 18 years.
4. Availability to meet the requirements of the protocol.
5. Negative Rapid Serological Test of SARS-CoV-2

Exclusion Criteria:

1. Previous SARS-CoV-2 infection
2. Pregnancy or breastfeeding.
3. Suspected of active viral or bacterial infection.
4. Symptoms compatible with COVID-19, despite a negative PCR test.
5. Vaccination in the last 4 weeks or planned vaccination during the study period, regardless of the type of vaccine.
6. Participation in a research that requires experimental intervention (does not include observational studies) in the previous month before signing the Consent or during the study.
7. Severely immunocompromised people. This exclusion category includes:

   1. Subjects with human immunodeficiency virus (HIV-1).
   2. Neutropenic subjects with less than 500 neutrophils / mm3.
   3. Subjects with solid organ transplantation.
   4. Subjects with bone marrow transplantation.
   5. Subjects undergoing chemotherapy.
   6. Subjects with primary immunodeficiency.
   7. Severe lymphopenia with less than 400 lymphocytes / mm3.
   8. Treatment with any anti-cytokine therapy.
   9. Oral treatment with steroids, defined as daily doses of 10 mg prednisone or equivalent for more than 3 months.
8. Malignancy, or active solid or non-solid lymphoma from the previous two years.
9. BCG vaccination in the last 10 years.
10. Treatment with Manremyc® for the last 6 months.
11. Chloroquine or hydroxychloroquine administration in the last two weeks.
12. Direct involvement in the design or execution of the MANRECOVID19 clinical trial.
13. Retirement, transfer, long-term leave (> 1 month) due to scheduled surgery or any other event that makes it impossible to work in person at your health center during the months following the recruitment to the study.
14. Employee at the health center <22 hours per week.
15. Do not have a smartphone.
16. Detection by the investigator of lack of knowledge or willingness to participate and comply with all requirements of the protocol.
17. Any other findings that, at the discretion of the investigator, may compromise compliance with the protocol or that may influence significantly the interpretation or the results of the effects of probiotic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Documented cumulative incidence of SARS-CoV-2 infection | up to 4 months
  % of positive serology at the end of the study or positive PCR test in the course of routine clinical practice

SECONDARY OUTCOMES:
Documented sick leave for SARS-CoV-2 | up to 4 months (cumulative)
  Number of days Documented as sick leave for SARS-CoV-2
days off work due to the quarantine | up to 4 months
  Number of days off work due to the quarantine imposed as a consequence to have acute respiratory symptoms, fever or infection documented by SARS-CoV-2
Quarantine imposed by close contact outside the center with SARS-CoV-2 positive | up to 4 months
  Number of days in quarantine imposed by close contact outside the center with SARS-CoV-2 positive
Fever | Up to 4 months
  Number of days of self-reported fever (≥38 ºC)
Cumulative incidence of self-reported acute respiratory symptoms | up to 4 months
  Cumulative incidence of self-reported acute respiratory symptoms
Number of days of self-reported acute respiratory symptoms | up to 4 months
  Number of days of self-reported acute respiratory symptoms
Incidence of pneumonia | up to 4 months
  Number of participants with pneumonia confirmed by X-ray
Cumulative incidence of death from documented SARS-CoV-2 infection | Up to 4 months
  Cumulative incidence of death from documented SARS-CoV-2 infection
Incidence of admission to ICU | Up to 4 months
  Cumulative incidence of admissions to intensive care unit for documented SARS-CoV-2 infection
Days in IUC | Up to 4 months
  Number of days admitted to the ICU for documented SARS-CoV-2 infection
Incidence of mechanical ventilation | Up to 4 months
  Cumulative incidence of need for mechanical ventilation due to documented SARS-CoV-2 infection
Incidence of hospital admissions | Up to 4 months
  Cumulative incidence of hospital admissions for documented SARS-CoV-2 infection
Days of hospitalization | Up to 4 months
  Number of days of hospitalization for documented SARS-CoV-2 infection
Levels of IgG | Up to 4 months
  Levels of IgG
Levels of IgM | Up to 4 months
  Levels of IgM
Levels of SARS-CoV-2 antibodies at the end of the study period | Up to 4 months
  Levels of SARS-CoV-2 antibodies at the end of the study period

OTHER OUTCOMES:
AEs | Up to 4 months
  All adverse events reported by the subjects, both serious and non-serious, will be collected. All events related to a SARS-CoV-2 infection will be exempted from collection, as they will be collected as part of the associated symptoms
SAEs | Up to 4 moths
  All thoseAdverse Events that lead to hospitalization of the patient, that endanger his life or cause or may cause death.

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - CAP Cornellà (La Gavarra), Cornellà de Llobregat, Barcelona
  - CAP Maresme, Mataró, Barcelona
  - Cap Sant Fèlix, Sabadell, Barcelona
  - EAP Riu Nord, Santa Coloma de Gramenet, BArcelona
  - Hospital Universitari Germans Trias i Pujol UBP Riscos Laborals, Badalona,, Badalona

IPD SHARING:
Plan to Share IPD: No